CLINICAL TRIAL: NCT03101813
Title: International Diffuse Intrinsic Pontine Glioma (DIPG)/Diffuse Midline Glioma (DMG) Registry and Repository
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The DIPG Collaborative (Unknown)
Responsible Party: Sponsor
Other Study IDs: DIPG/DMG-REGISTRY-REPOSITORY
Record Dates: First submitted 2017-03-08; First posted 2017-04-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant; Diffuse Midline Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Sources of tumor tissue may be from diagnostic biopsy, surgery or autopsy samples. Fresh tumor tissue may be utilized immediately for biological studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Doctors and other medical scientists want learn about the biology of DIPG/DMG and to develop better ways to diagnose and treat patients with DIPG/DMG. To do this, they need more information about the characteristics of DIPG/DMG tumors. Therefore, they want to establish a central location for clinical information and tumor tissue collected from DIPG/DMG patients.

The purposes of this study are:

* To enroll patients diagnosed with DIPG/DMG in the International DIPG/DMG Registry and Repository.
* To provide a central location for clinical information, scans, and tissue samples from patients with DIPG/DMG enrolled in the registry.
* To collect tissue samples in order to study how DIPG/DMG works on the molecular level. Researchers may use the tissue samples to study molecules such as proteins and DNA. Proteins are needed for the body to function properly and DNA is the molecule that carries our genetic information. Other researchers will be able to use the stored samples in the future to learn more about DIPG/DMG. The information researchers get from the research studies will be kept in the registry along with the clinical information.
* To help investigators around the world to work together to make more consistent diagnosis and better design of future research studies. We hope this will lead to better treatments for DIPG/DMG in the future.

DETAILED DESCRIPTION:
There are limited data regarding the biology of diffuse intrinsic pontine gliomas (DIPG) and diffuse midline gliomas (DMG). This project provides the infrastructure for acquisition of biological specimens, imaging, and correlative clinical data to facilitate biology studies in this group of patients. The goal of the DIPG/DMG registry is to promote collaborations amongst investigators to allow timely data and/or specimen dissemination for future research studies and to develop classification systems, uniform standards of diagnosis, assessment and response, ultimately leading to the development of effective therapies for children with DIPG/DMG.

This registry will collect clinical, demographic, radiological and pathological data and specimens (if available) from patients with DIPG/DMG, both prospectively (in newly diagnosed or currently living patients), as well as retrospectively (in patients who are deceased). Cases are identified through:

1. Existing clinical and/or cancer registry databases
2. Referrals from clinicians, surgeons, or pathologists
3. Families initiating contact with Registry staff directly

The following data/materials will be collected:

Clinical: Demographic data, date of diagnosis, signs and symptoms at diagnosis, laboratory data, detailed treatment data (e.g. types and dates of surgeries (if any), chemotherapy, radiotherapy), best response to treatment, dates of progression, types of progression (local or metastatic), and follow-up data.

Imaging: All radiographic imaging obtained since diagnosis will be requested at the time of study entry.

Pathology Central Review: If glass slides (stained or unstained) or paraffin blocks of tumor tissue (from biopsy or autopsy) are available, they will be requested at the time of registry entry but are not mandatory for enrollment.

Bioinformatics repository: Collection of existing molecular and/or genomic data or analysis that has been performed as well as prospective analysis of tissue from the registry will be submitted to a central bioinformatics repository and may be linked to clinical data housed in the DIPG/DMG registry.

Tissue Collection and Storage for Future Research: If available, participants' frozen tissue may be submitted for banking and future research.

Data stored in the Registry may be used to provide statistical data for scientific presentations and for preparation of peer-reviewed manuscripts. No personal data can be traced to the study manuscripts or presentations. Data and specimens will be released for research proposals upon approval from the International DIPG/DMG Registry Committee.

The International DIPG/DMG Registry and Repository is not associated with any oncology group cooperative study or treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients of any age (living or deceased) with a diagnosis (either current or past) of a DIPG/DMG tumor
* Unless the patient is deceased, all patients and/or one parent or legal guardian must provide written informed consent as well as HIPAA/release of information consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of any age (living or deceased) with a diagnosis (either current or past) of a DIPG/DMG tumor.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2037-06 (Estimated); Study Completion 2047-06 (Estimated)

PRIMARY OUTCOMES:
Identify the biological factors contributing to DIPG/DMG | Through study completion, anticipated to be 25 years
  To implement a central repository for clinical, radiological, pathological and demographic data and specimens from patients with DIPG.

SECONDARY OUTCOMES:
Identify genetic and molecular signature of diffuse intrinsic pontine gliomas and diffuse midline gliomas. | Through study completion, anticipated to be 25 years
  correlate registry data to a bioinformatics repository of molecular data on DIPG/DMG
Identify radiographic characteristics of DIPG/DMG | Through study completion, anticipated to be 25 years
  develop classification systems, uniform standards of diagnosis, assessment and response

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Hoffman, DO, Study Chair — Phoenix Children's Hospital; Trent Hummel, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical, radiographic, pathologic, genomic data and biological specimens may be released to qualified investigators after a subset of the study committee for this protocol has judged their proposals for scientific merit, clinical priority, and feasibility.
  Patient-identifying data/specimens will never be released to investigators. If the use of the samples and/or data released from the repository constitutes human subjects research per 45 CFR 46 or genetic research, IRB approval will be required to be submitted with the investigator's application.

REFERENCES:
- See also: International DIPG Registry and Repository website — http://dipgregistry.org/